CLINICAL TRIAL: NCT04905225
Title: The Gender Specific Effect on the Results of Ascending Aortic Replacement in Small Ascending Aortic Aneurysm
Brief Title: The Gender Specific Effect on the Results of Ascending Aortic Replacement
Status: Completed | Type: Observational
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: Tomsk NRMC CRI
Record Dates: First submitted 2021-05-23; First posted 2021-05-27 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Ascending Aortic Aneurysm
MeSH Terms: conditions — Aneurysm, Ascending Aorta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ascending aortic replacement: Ascending aortic replacement in ascending aortic aneurysm in men and women
  Interventions: Procedure: Ascending aortic replacement

INTERVENTIONS:
Procedure: Ascending aortic replacement — Surgical access will be performed through a median sternotomy. Ascending aortic repair is performed under conditions of cardiopulmonary bypass (CPB) and MHCA with unilateral ACP via innominate artery with a flow rate of 8-10 ml/kg/min and perfusion pressure of 60-80 mmHg. Once CPB is instituted, the aortic cross-clamp is applied, and the heart is arrested with antegrade cardioplegia. Hemiarch replacement involves resection lesser curve of the aortic arch from the base of the innominate artery (Zone 0) to a point immediately distal to the nadir of the lesser curvature (Zone 3 or Zone 2 if the left subclavian artery was too far).

SUMMARY:
The aim of our study is to analyze the early and late results in men and women who underwent ascending aortic replacement in antegrade cerebral perfusion (ACP) with mild-to-moderate hypothermic circulatory arrest. Female gender is associated with poorer outcomes after surgical aorta replacement. Data on gender specific differences after ascending aortic replacement are conflicting.

DETAILED DESCRIPTION:
Description of the procedures:

All surgical procedures will be performed via median sternotomy. During the aortic arch anastomosis, continuous, unilateral SACP using innominate artery will be employed. Unilateral SACP may be converted to bilateral ACP at the surgeon's discretion if adequate cerebral flows are not achieved or if there are concerns with cerebral oximetry measurements.

Once on CPB, the patient will be cooled to a nasopharyngeal (NP) temperature of either 26-32 °C. Rectal temperature with be monitored as an additional temperature sites. Unilateral SACP will only be initiated once the target temperature has been reached. SACP via the innominate artery will be commenced with target flows of 8-10 ml/kg/min and perfusion pressure of 60-80 mmHg. Perfusion adequacy will be evaluated using measurement of blood pressure in both radial arteries and cerebral oximetry using near-infrared spectroscopy (NIRS).

After completion of the aortic hemiarch replacement, CPB will be resumed and the patient re-warmed to 36 °C prior to coming off CPB, with a = 1 °C temperature difference between temperature monitoring sites (NP and rectal).

Intraoperative information will be collected from the anesthetic record, surgical notes and perfusion records. Intraoperative data collection will include total operative time, CPB time, cross-clamp time, hypothermic cardiac arrest time, uSACP time, lowest nasopharyngeal and rectal temperature, arterial pressure in both radial arteries, perfusion rate and perfusion pressure during both of CPB and unilateral SACP, lowest hemoglobin concentration (g/L) and hematocrit (%), acid-base indices, intraoperative red blood cell transfusion (units), highest dose/agent used for intraoperative inotrope or vasopressor support. Also during the surgery will be performed NIRS and BIS-monitoring(bispectral index).

Postoperative data will include valuation of following indicators: mortality (hospital mortality and death from any cause); neurological injury (TIA, stroke, delirium), MRI and CT-scan only in event of postoperative stroke; acute kidney injury (creatinine level prior and 1, 2, 4 postoperative day (POD), renal replacement therapy (dialysis); time of mechanical ventilation; re-exploration for bleeding, tamponade or other reasons; postoperative transfusion (packed red blood cells, platelets, fresh frozen platelets, cryoprecipitate); postoperative myocardial infarction (electrocardiogram and troponins); length of stay (intensive care unit and total hospital days).

Follow-up information will be collected using direct or phone contact with patients, relatives, or physicians.

ELIGIBILITY:
Inclusion Criteria:

* Patients with small ascending aortic aneurysm (5.0-5.5 cm)
* Elective procedure
* Able to provide written informed consent

Exclusion Criteria:

* Surgery for acute aortic dissection or emergent operations
* Refusal of surgical treatment
* Oncological disease (high degrees)
* Multiple organ failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ascending aortic aneurysm with Hemiarch replacement
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Operative mortality | During the first 30 days after the procedure
  Operative mortality (%) as assessed by data linkage to medical records Comparison of men vs women in aortic hemiarch surgery with respect to the incidence of death
All-cause mortality | Up to 5 years
  all-cause mortality as assessed by data linkage to medical records or or phone contact with relatives or physicians

SECONDARY OUTCOMES:
Perioperative Myocardial Infarction | During the first 30 days after the procedure (assessed by daily serum assay and ECG in the ICU and every 5 days after discharge from ICU. )
  Incidence of the myocardial infarction (%) is assessed by complex evaluation based on the ECG and echocardiographic changes as well as increase of the troponin level using serum assay
Rates of re-exploration for bleeding | During the first 3 days after the procedure
  Percentage of patients requiring re-exploration for bleeding.
Respiratory failure | During the first 30 days after the procedure
  Percentage of patients requiring prolonged lung ventilation (> 72 hours) or tracheostomy
The duration of a patient's stay in the intensive care unit and on the hospital ward | Up to 90 days after surgery
  The duration of a patient's stay in the intensive care unit and on the hospital ward
Incidence of Acute Kidney Injury (AKI) | During the first 30 days after the procedure
  Percentage of patients requiring renal replacement therapy (i.e. haemodialysis or haemofiltration
Composite of neurologic injury | During the first 30 days after the procedure
  Percentage of patients with neurological complications is assessed. Single assessment by CT or MRI. More often if necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Boris N Kozlov, Dr, Study Director — TOMSK NRMC CARDIOLOGY RESEARCH INSTITUTE
Locations (1):
- Tomsk NRMC, Tomsk, Russia